CLINICAL TRIAL: NCT05268393
Title: Feasibility Trial of a Mindfulness Based Intervention in Youth With Type 1
Brief Title: Feasibility Trial of a Mindfulness Based Intervention in Youth With Type 1 Diabetes
Acronym: BREATHE-T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Eleanor Mackey, Associate Professor, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15464; R34AT011035 (NIH)
Record Dates: First submitted 2022-02-15; First posted 2022-03-07 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: type1diabetes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BREATHE-T1D (Experimental): BREATHE-T1D is a 6-week group mindfulness program adapted specifically for teens with type 1 diabetes.
  Interventions: Behavioral: BREATHE-T1D
- BREATHE-T1D Health Education (Placebo Comparator): The health education placebo comparator is a 6-week group diabetes-specific education program designed to be informational but not supportive.
  Interventions: Behavioral: BREATHE-T1D

INTERVENTIONS:
Behavioral: BREATHE-T1D — BREATHE-T1D is a mindfulness based intervention adapted from Learning to BREATHE specifically for teens with type 1 diabetes.

SUMMARY:
Type 1 diabetes (T1D) is one of the most common chronic illnesses of childhood. The involved treatment regimen, including daily insulin administration/pump management, frequent blood glucose checks, and careful track-ing of food intake, places a high-stress burden on patients and their families. Adolescence is a particularly risky time for T1D management given a marked decline in treatment adherence and glycemic control. Over 80% of adolescents with T1D have poor glycemic control (A1c >7.5%), and one significant risk factor is the increase in negative affectivity, including depression and anxiety symptoms, that distinguish adolescents with T1D. Elevated depression and anxiety symptoms affect 40% of teens with T1D. Preliminary data support the notion that negative affectivity contributes to diminished treatment adherence and worsening of glycemic control, partially through the effects of negative affectivity on stress-related behavior such as maladaptive eating behavior (e.g., dietary restriction, uncontrolled eating patterns, and insulin omission for weight control). There is no gold-standard approach to address the poor glycemic control seen in adolescents with T1D. The creation of novel, targeted interventions, tailored for the developmental needs of adolescents with T1D and the particular burdens of coping with their chronic illness, are needed. Mindfulness-based interventions delivered to adolescents without T1D, including the team's preliminary work in teens with depression and weight-related disorders, have shown promise in treating negative affectivity, maladaptive eating behavior, and health outcomes. A mindfulness-based approach may be well-suited for adolescents with T1D, but given that the mechanisms of association among negative affectivity, stress-related behavior, and self-care are unique to individuals with T1D, interventions must be specifically tailored for this population. The goal of this study is to, therefore, adapt an existing 6-session mindfulness-based intervention, Learning to BREATHE, for use with adolescents with T1D (BREATHE-T1D). The first specific aim of the study is to adapt BREATHE for adolescents with T1D and to adapt a relevant and credible health education comparison curriculum (HealthEd-T1D). The second aim is to carry out a 2-way pilot randomized controlled trial to evaluate the feasibility and acceptability of BREATHE-T1D and HealthEd-T1D. The result of the current study will be a feasible and acceptable mindfulness intervention and comparison curriculum that can be evaluated in an efficacy trial. The multidisciplinary study team contributes complementary areas of expertise in adolescents with T1D, behavioral intervention development, negative affectivity and maladaptive eating behavior, adolescent mindfulness-based intervention, qualitative data analysis, and delivery of behavioral health interventions via telehealth. The study's innovative approach will enable the investigators to establish a feasible/acceptable intervention tailored for adolescents with T1D, leading to a future proposal for a full-scale efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* age 12-17y
* T1D, with at least 1-year duration of illness
* negative affectivity, defined as clinically elevated scores (T-score >55 indicating at least mild depression/anxiety symptoms on either the PROMIS short form-depression and/or anxiety scales)
* A1c >7.5%
* English-speaking

Exclusion Criteria:

* no cognitive or developmental delays which would interfere with their ability to participate in the study
* are able and willing to complete questionnaires and intervention via the internet
* do not have severe depression or active or recent (within the past two months) suicidal ideation
* have no other serious medical conditions (e.g., cystic fibrosis, cancer).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lupini F, Basch M, Cooke F, Vagadori J, Gutierrez-Colina A, Kelly KP, Streisand R, Shomaker L, Mackey ER. BREATHE-T1D: Using iterative mixed methods to adapt a mindfulness-based intervention for adolescents with type 1 diabetes: Design and development. Contemp Clin Trials. 2024 Jul;142:107551. doi: 10.1016/j.cct.2024.107551. Epub 2024 Apr 29. PMID 38692428
- [Result] Basch M, Lupini F, Ho S, Dagnachew M, Gutierrez-Colina AM, Patterson Kelly K, Shomaker L, Streisand R, Vagadori J, Mackey E. Mindfulness-based group intervention for adolescents with type 1 diabetes: initial findings from a pilot and feasibility randomized controlled trial. J Pediatr Psychol. 2024 Oct 1;49(10):769-779. doi: 10.1093/jpepsy/jsae071. PMID 39212647

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Started | 20 | 22
Completed | 18 | 21
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (1.8) | 14.7 (1.9) | 14.8 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 6 | 11
  White | 10 | 9 | 19
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42
HbA1c [Mean (Standard Deviation); unit: percentage] — HbA1c was abstracted from medical records and assessed at clinic visits. Optimal HbA1c value is <7.0%. Lower values represent more optimal glycemic control.
  percentage | 7.7 (1.1) | 8.7 (2.5) | 8.2 (2.0)
Depression [Mean (Standard Deviation); unit: T-score] — The PROMIS self-report brief depression measure uses t-scores with scores >55 indicative of depressive symptoms. Higher scores indicate more depressive symptoms. T-scores can be interpreted as 50 indicating the population mean with a standard deviation of 10.
  T-score | 58.5 (9.0) | 56.2 (8.7) | 56.7 (8.6)
Anxiety [Mean (Standard Deviation); unit: T-score] — The PROMIS self-report brief anxiety measure uses t-scores with >55 indicating significant anxiety symptoms and higher scores indicating greater levels of anxiety. T-scores can be interpreted as 50 indicating the population mean with a standard deviation of 10.
  T-score | 58.8 (7.9) | 57.1 (7.2) | 57.6 (7.6)
Disordered Eating [Mean (Standard Deviation); unit: units on a scale] — The Diabetes Eating Problems Survey Revised (DEPS-R) is a measure of disordered eating behavior in individuals with type 1 diabetes, consisting of 16 items. Adolescents are asked to rate how often they agree or engage in each behavior, on a six-point Likert scale (ranging from never to always), with higher scores indicating greater severity of disordered eating behaviors. Total scores can range from 0-80. A score of ≥20 is considered clinically significant, as it has been correlated with poorer glycemic control and potential increased risk of diabetes complications.
  units on a scale | 21.8 (11.1) | 23.4 (15.3) | 22.6 (13.3)
Diabetes Distress [Mean (Standard Deviation); unit: units on a scale] — The Problem Areas in Diabetes-Teen (PAID-T) is a 14-item measure of diabetes distress in adolescents with type 1 diabetes. Adolescents are asked how often each diabetes-related problem applied to them in the past month, on a six-point Likert scale (ranging from not a problem to serious problem), with higher scores indicating greater severity and a clinical cutoff of >44.
  units on a scale | 61.7 (23.5) | 60.1 (21.9) | 60.9 (22.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Enrolled of Eligible Participants Screened
Description: The percentage is calculated first by identifying the number of enrolled participants divided by eligible participants. 42 total patients were eligible once screened across the 10 month enrollment period. 42 total then enrolled in the study.
Time Frame: During screening (10 months total)
Population: Number of participants screened (42 in all across 10 months were eligible for the study following screening).
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants prior to randomization.
Arm/Group | All Participants
Number analyzed (Participants) | 42
Participants | 42

2. Primary Outcome: Number of Weeks to Enroll Participants to Form One Cohort
Description: Number of weeks to enroll 10 participants to be randomized 5 per group
Time Frame: During screening (10 months)
Population: All randomized participants
Measure: Mean (Full Range); unit: weeks
Groups:
- All Participants: Participants were recruited in cohorts (groups of 10) and then were randomized within cohort to each of the two programs.
Arm/Group | All Participants
Number analyzed (Participants) | 42
weeks | 8 [5 to 10]

3. Primary Outcome: Percentage of Participants With Data Collected
Description: Number of participants with data at each time point.
Time Frame: Baseline, Immediate post-intervention (2-3 months post baseline), 3 month follow up (5-6 months post baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 20 | 22
Participants
  Immediate follow up | 18 | 21
  3 month follow up | 18 | 21

4. Primary Outcome: Percentage of Attended Sessions
Description: Number of intervention sessions (calculated by multiplying number of expected sessions by number of participants for total possible sessions held) attended divided by total number of intervention sessions expected per group.
Time Frame: Immediate post-intervention follow-up (2-3 months post baseline)
Population: The aim was for each participant to attend 6 program sessions. Therefore, the number of expected sessions multiplied by the number of participants are reflected in the overall number of units analyzed.
Measure: Number; unit: percentage of sessions attended overall
Units Other Than Participants: Sessions
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 18 | 21
Number analyzed (Sessions) | 108 | 126
percentage of sessions attended overall | 99 | 100

5. Primary Outcome: Satisfaction With Intervention Program
Description: Satisfaction report by participants
Time Frame: Immediate post-intervention follow-up (2-3 months post-baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 18 | 21
Participants | 15 | 19

6. Secondary Outcome: Mindful Attention Awareness Scale
Description: Assessed via teen report. Scores are calculated as an average score of all items with a range of 1 (minimum) to 6 (maximum) with higher scores indicating more mindful attention in daily life.
Time Frame: Baseline, Immediate post-intervention (2-3 months post baseline), 3 month follow up (5-6 months post baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 16 | 21
score on a scale
  Immediate follow up | 3.8 (.87) | 3.8 (.99)
  3 month follow up | 3.9 (1.3) | 3.9 (1.0)

7. Secondary Outcome: Five-Facet Mindfulness Questionnaire
Description: Assessed via teen report. Scores are calculated as a total score across all items in the scale with a range of 1 (minimum) to 5 (maximum) and total scores presented are a sum of the sub scale (observing, describing, acting with awareness, nonjudging, and non-reactivity) with possible scores ranging from 5-25 with higher scores indicating more mindfulness.
Time Frame: Baseline, Immediate post-intervention follow up (2-3 months post baseline), 3 month follow up (5-6 months post-baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 16 | 21
score on a scale
  Immediate follow up | 19.4 (2.2) | 18.5 (3.3)
  3 month follow up | 19.9 (2.9) | 19.1 (3.7)

8. Secondary Outcome: PROMIS Depression Short Form - Adolescent Report
Description: Scores are calculated as t-scores with higher scores indicating more depressive symptoms. T-scores (range 0-100) over 55 indicate clinically significant depressive symptoms. Interpretation of t-scores is based on a mean of 50 and standard deviation of 10.
Time Frame: Baseline, Immediate post-intervention follow up (2-3 months post baseline), 3 month follow up (5-6 months post baseline)
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 18 | 21
t-score
  Immediate follow up | 55.9 (9.4) | 54.8 (9.8)
  3 month follow up | 53.0 (9.6) | 56.0 (9.2)

9. Secondary Outcome: PROMIS Anxiety Short Form - Adolescent Report
Description: Scores are calculated as t-scores (range 0-100) with higher scores indicating more anxiety symptoms.T-scores over 55 indicate clinically significant anxiety symptoms. Interpretation of t-scores is based on a mean of 50 and standard deviation of 10.
Time Frame: Baseline, Immediate post-intervention (2-3 months post baseline), 3 month follow up (5-6 months post baseline)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 18 | 21
T-score
  Immediate follow up | 56.7 (6.6) | 53.8 (8.1)
  3 month follow up | 53.8 (7.6) | 54.0 (8.6)

10. Secondary Outcome: Diabetes Eating Problems Survey Revised
Description: Teen report with higher scores indicating more disordered eating behaviors with scores over 25 indicating clinically significant problems. Total scores range from 0 to 64 with higher scores indicating more disordered eating behaviors.
Time Frame: Baseline, Immediate post-intervention (2-3 months post baseline), 3 month follow up (5-6 months post baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 18 | 21
score on a scale
  Immediate follow up | 18.6 (13.1) | 18.2 (14.2)
  3 month follow up | 19.3 (13.1) | 20.0 (16.5)

11. Secondary Outcome: UPPS-P Negative Urgency Subscale
Description: Teen report on the UPPS-P Negative Urgency subscale with higher scores indicating more likelihood to act impulsively when experiencing a negative mood. Scores are calculated with an average which can range from 1(minimum) to 4 (maximum).
Time Frame: Baseline, Immediate post-intervention (2-3 months post baseline), 3 month follow up (5-6 months post baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 17 | 20
score on a scale
  Immediate follow up | 2.52 (.85) | 2.42 (.68)
  3 month follow up | 2.65 (.58) | 2.64 (.63)

12. Secondary Outcome: Self-Care Inventory
Description: Teen report on the Self-Care Inventory, a measure of diabetes management with higher scores indicating better self-care for diabetes. Average scores range from 1 (minimum) to 5 (maximum).
Time Frame: Baseline, Immediate post-intervention (2-3 months post baseline), 3 month follow up (5-6 months post baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 17 | 20
units on a scale
  Immediate follow up | 3.73 (.66) | 3.53 (.77)
  3 month follow up | 3.68 (.71) | 3.48 (.76)

13. Secondary Outcome: Problem Areas in Diabetes - Teen
Description: The Problem Areas in Diabetes-Teen (PAID-T) is a 14-item measure of diabetes distress in adolescents with type 1 diabetes. Adolescents are asked how often each diabetes-related problem applied to them in the past month, on a six-point Likert scale (ranging from not a problem to serious problem), with scores reflecting a total across 14 items and higher scores indicating greater severity and a clinical cutoff of >44. Scores can range from 14-84.
Time Frame: Baseline, immediate post intervention (2-3 months post baseline), 3 month follow up (5-6 months post baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 18 | 21
score on a scale
  Immediate follow up | 49.8 (22.4) | 53.1 (22.7)
  3 month follow up | 46.8 (19.4) | 49.1 (21.1)

14. Secondary Outcome: Glycemic Control
Description: HbA1c is a measure of an average blood glucose level over the past 3 months and will be abstracted from the medical record as it is assessed at each regular diabetes clinic visit. HbA1c typically ranges from 4% to >14%.
Time Frame: Baseline, immediate post intervention follow up (2-3 months post baseline), 3 month follow up (5-6 months post baseline)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 16 | 16
percentage
  Immediate follow up | 7.95 (1.3) | 8.79 (2.5)
  3 month follow up | 7.6 (1.0) | 8.7 (2.6)

15. Secondary Outcome: Interventionist Adherence to Session Manuals
Description: Supervisors listened to recordings of sessions for both programs and completed checklists assessing for the number of expected intervention components included in the sessions. Therefore, values reflect the percentage of expected intervention components included across all program sessions calculated at the end of the intervention period (week 6) for each group cohort.
Time Frame: Week 6 of intervention
Population: All participants were included as these were ratings of sessions, not individual by participant.
Measure: Mean (Standard Deviation); unit: percentage of intervention components
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
Number analyzed (Participants) | 20 | 22
percentage of intervention components | 100 (0) | 100 (0)

ADVERSE EVENTS:
Time Frame: Screening through 3 month follow up, an average of 6 months.
Arm/Group | BREATHE-T1D | BREATHE-T1D Health Education
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/21
Other Adverse Events (participants affected / at risk) | 0/18 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT05268393/Prot_SAP_000.pdf